CLINICAL TRIAL: NCT01285947
Title: A Pilot Study of 20 Subjects: Pain Experience in Naive vs. Non-naive Subjects Undergoing Energy-based Dermatologic Procedures
Brief Title: Comparing the Pain Experience Between Patients Who Have and Who Have Not Undergone Dermatologic Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Associate Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STU 40788
Record Dates: First submitted 2011-01-27; First posted 2011-01-28 (Estimated); Results first posted 2014-02-05 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Pain
Keywords: pain experience; energy devices; Ulthera; Thermage; VBeam
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naive Subjects (Other): Subjects who have not previously undergone energy-based dermatologic procedures in the past.
  Interventions: Device: Thermage; Other: Needle Application; Device: VBeam Laser; Device: Ulthera
- Non-Naive Subjects (Other): Subjects who have previously undergone energy-based dermatologic procedures in the past.
  Interventions: Device: Thermage; Other: Needle Application; Device: VBeam Laser; Device: Ulthera

INTERVENTIONS:
Device: Thermage — Radiofrequency Device - specific setting will be determined by the location and thickness of skin. Periorbital: 58-140 J/cm2 Midface: 81-124 J/cm2 Abdomen: 95-181 J/cm
Other: Needle Application — 30-gauge needle insertion into skin
Device: VBeam Laser — Pulsed Dye Laser at the following settings: 7.5 J, 0.6ms, 10mm, DCD 30/20
Device: Ulthera — Ultrasound Device at the following settings:
  Transducer Frequency Depth Image Depth DS 7-3.0 7 MHz 3.0mm 0-8mm DS 4-4.5 4 MHz 4.5mm 0-8mm DS 7-4.5 7 MHz 4.5mm 0-8mm

SUMMARY:
The purpose of this study is to compare the pain experience of patients who have not had dermatologic procedures (previously "unexposed") using energy devices (lasers, radiofrequency, ultrasound, etc.) with patients who have previously had procedures (previously "exposed") using energy devices. Based on previous clinical encounters, individuals with no prior experience with cosmetic procedures appear to experience more pain. However, no study to date has thoroughly examined this observation. As a result, this study has been designed to find a possible difference in pain perception between previously exposed and unexposed patients undergoing cosmetic procedures using energy devices.

DETAILED DESCRIPTION:
Twenty subjects will be enrolled in the study: 10 subjects who have had cosmetic procedures in the past and 10 subjects who have not had such procedures. For each subject, pain tolerance in three areas will be assessed: temple, midface/cheek, and abdomen. In two areas of the face (temple and midface/cheek), a small sterile needle will be inserted into the skin along with three applications of the following devices that are FDA approved for use on the face: an ultrasound device (Ulthera), a pulsed dye laser (VBeam), and a radiofrequency (Thermage) device. Additionally, the abdomen will receive three of these four devices in a randomized order: small sterile needle insertion, a pulsed dye laser (VBeam) pulse, and a radiofrequency (Thermage) exposure (the ultrasound device, Ulthera, will not be used on the abdomen because it is currently not FDA approved for this indication). Subjects will then be asked to rate their pain after each application at each individual site using a pain scale. In addition, subjects will complete a questionnaire regarding their pain experiences and other possibly related factors before and after the procedures.

ELIGIBILITY:
Inclusion Criteria

1. Subjects of both genders, 18 to 65 years of age.
2. Subjects who are in good health.
3. Non-naïve (patients who have not had cosmetic procedures using energy devices): Subjects who have had three or more non-ablative laser procedures or any skin tightening procedure using an energy device.
4. Subjects who understand and are willing to provide informed consent for participation in the study and are able to communicate with the investigator.

Exclusion Criteria:

1. Subjects who have an active skin disease or skin infection in or around the treatment.
2. Subjects who are unable to understand the protocol or give informed consent.
3. Subjects with photophobia or who are unable to tolerate the treatments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naive Subjects | Non-Naive Subjects
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naive Subjects | Non-Naive Subjects | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Pain Rated by Subjects
Description: The mean pain scores will be compared between naïve subjects and non-naïve subjects averaged over the anatomical sites: periocular (temple), midface/cheek, and abdomen and over all the different treatments.
  Pain scores were recorded along a Visual Analog Scale (VAS) with 0 (no pain- better) to 10 (maximal pain-worst). This is a 10 cm long line in which the subject was asked to draw a line on the scale with 0 (no pain- better) at one end to 10 (maximal pain-worst) at the other end. The drawn line was measured on the 10 cm line using a ruler to obtain the score.
Time Frame: 3 hours for all treatments in one visit
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Naive Subjects | Non-Naive Subjects
Number analyzed (Participants) | 10 | 10
Units on a scale | 2.3 (1) | 2.2 (1.4)

ADVERSE EVENTS:
Arm/Group | Naive Subjects | Non-Naive Subjects
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes